CLINICAL TRIAL: NCT01755065
Title: Clinical Meaning of Visual Analog Scales (VAS) for Teenage Pediatric Patients Undergoing Laparoscopic Surgical Procedures
Brief Title: Clinical Meaning of Visual Analog Scales(VAS) for Teenage Pediatric Patients Undergoing Laparoscopic Surgical Procedures
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Mihaela Visoiu, Assistant Professor of Anesthesiology, University of Pittsburgh
Other Study IDs: PRO12020593
Record Dates: First submitted 2012-12-19; First posted 2012-12-21 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2015-04

CONDITIONS: Postoperative Pain
Keywords: laparoscopic surgery; teenager
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Teenager laparoscopic patients

SUMMARY:
The purpose of this study is to find a more accurate postoperative pain assessment for teenager patients. This is important because a patient should not have a very strong pain medication such as morphine if the pain is just mild.

DETAILED DESCRIPTION:
Pain is a sensory and emotional experience, modified by multiple factors, including meaning, context, previous pain experience, culture, gender, expectation, anxiety, depression, fear, family and social factors. Hospitalized teenager patients (11-18 years) admitted to surgical services experience high prevalence of moderate and severe pain.1 The VAS (Visual Analog Scale, 0 mm "no pain", to 100 mm," the worst pain possible ") is used to assess postoperative pain for teenager patients. The reliability and validity of this scale was proven but clinical significance of VAS pain score is not clear. 2 There is an increased focus on very good pain control and is a common practice that patients with moderate or severe pain scores (numeric rating score, more than 4) to receive opioid pain medication 3, regardless of pain behavior or health care providers' input , and this can result in various side effects. Pediatric nurses administer more pain medications to the children who vocalize their pain. 4 Numerous clinical trials of postoperative pain treatment in teenager use only VAS pain scores to assess the effectiveness of a studied pain medication.

Although the treatment of pain may be a basic human right, that does not mean that all teenager patients require opioids administration if they report high pain scores. It is our observation that teenager's pain behavior does not always correlate with the magnitude of reported pain scores by the patient and different caregivers. Concomitant parental and nurse observation of teenager's pain behavior can provide additional information about pain severity. Minimal correlation between VAS pain scores reported by teenager and caregivers does not mean that pain severity is "unreal". Perioperative teenager's pain catastrophizing thoughts about pain, anxiety, and mood level can influence teenager's postoperative pain scores.

The authors aim is to develop a multi-modal assessment of postoperative pain for the teenager patient, using VAS pain scores reported by the teenager, nurse, and parent in association with the teenager's postoperative pain behavior, pain catastrophizing thinking, anxiety, and mood level. The subjects included in this study will be 206 teenager patients (11-17 years old) undergoing any laparoscopic surgical procedures. On postoperative day 1, the teenager will complete the following questionnaires: Visual Analog Scale from teenager (VAS teen), State-Trait Anxiety Inventory for Children (STAIC S - Anxiety), Pain Catastrophizing Scale for Children (PCS-C) and Brief Mood Introspection Scale (BMIS). The nurse taking care of the patient and one parent, preferable the mother, will complete the following questionnaires: Visual Analog Scale from parent (VAS p), Visual Analog Scale from nurse (VAS n), and Adolescent Pain Behavior Questionnaire from parent (APBQ-p), Adolescent Pain Behavior Questionnaire from nurse (APBQ-n). The main goal is to determine if VAS score reported by the teenager correlates with VAS scores reported by the parent and nurse, and with pain behavior scores reported by the nurse and family. Expected correlation is minimal (0.23-0.29) to moderate (0.3-0.49). Our second goal is to determine whether postoperative pain is associated with psychosocial factors such as teenager catastrophizing attention to pain, anxiety, and mood level. Expected correlation between postoperative VAS teen and teenager catastrophizing attention to pain, anxiety, and mood level is moderate (0.3-0.49) to high (>/=0.5).

To our knowledge, this is the first study to investigate all these variables together to assess postoperative pain for a teenager patient. The findings of this study may influence the medical decisions regarding administration of pain medication, allow for a safer and more effective use of opioids in postoperative period and would be very helpful for clinical and research practice.

ELIGIBILITY:
Inclusion Criteria:

* 11-17 years old, both male and female
* the patient is having any laparoscopic surgeries, elective or emergent, including robotic surgeries
* the patient will be admitted in hospital for at least 23 hours

Exclusion Criteria:

* Patient and family refusal
* Patient already enrolled in another study
* Non English-speaking patients and families
* Cognitive impairment
* Developmental delay
* Patients who experienced surgical, anesthesia or medical complications;
* Patients with chronic pain condition (pain more than 3 months)
* Patients medicated at home or in hospital with long acting opioid pain medication (methadone, oxycontin, oxymorphone ER, morphine slow release)
* Patients with psychiatric medical history (except attention deficit disorders such us: ADD and ADHD)
* Patients taking at home the following medication: clonidine, antipsychotic, antidepressant and anxiolytic medications.
* Patients taking drugs, including smoking marijuana and other recreational drugs
* Positive pregnancy test
* Laparoscopic surgical procedures converted to open procedures
* Patients will be discharged on the day of surgery.
* If none of the patient's parent will stay with the child during hospital stay, the patient will be not enrolled in the study. If all 8 questionnaires cannot be filled on the day after surgery, the patient will be discontinued from this study.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The participants will be selected based on medical records review and medical interview on the day of surgery: we plan to enroll 206 teenager patients (11-17 years old) with anticipated postoperative pain after any laparoscopic procedure and their parents and nurses.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2012-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Post-op pain score | 1 day post-operation

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States